CLINICAL TRIAL: NCT04765618
Title: The Incidence of Gall Stones After Bariatric Surgery and Its Association With Weight Loss
Status: Completed | Type: Observational
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Mahmoud alazawy, general surgery assistant lecturer, Helwan University
Other Study IDs: Helwan university
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: The Incidence of Gall Stones After Bariatric Surgery and Its Association With Weight Loss
Keywords: gall stones; ,bariatric surgery
MeSH Terms: conditions — Gallstones | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Procedure: bariatric surgery — laparoscopic sleeve gastrectomy,or gastric bypass

SUMMARY:
The incidence of Gall Stones after Bariatric surgery and its association with weight loss

DETAILED DESCRIPTION:
Gallstone (GS) formation is common in obese patients, particularly during rapid weight loss.This study aimed to determine the incidence of GS in patients underwent bariatric surgery (BS) and the influence of weight loss on GS formation.

ELIGIBILITY:
Inclusion Criteria:

* (BMI) ≥35kg/m2 with one or more obesity-related comorbidities
* a BMI > 40 kg/m2 without coexisting medical problems

Exclusion Criteria:

-a conrtaindication for bariatric surgery

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Methods This was a prospective study conducted in Helwan University Hospitals in Egypt including 148 consecutive patients underwent BS during the period between December 2018 and December 2019. Patients with preoperative negative abdominal ultrasound(US) for GS were followed-up for at least 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2018-12-26 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2020-12-26 (Actual)

PRIMARY OUTCOMES:
The incidence of Gall Stones after Bariatric surgery | the period between December 2018 and December 2019

SECONDARY OUTCOMES:
effect of weight loss on Gall Stones formation after Bariatric surgery | the period between December 2018 and December 2019
  effect of excess weight loss on gall stones formation after bariatric surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Dr.hossam hoseiny, Helwan, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Undecided: It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Talha A, Abdelbaki T, Farouk A, Hasouna E, Azzam E, Shehata G. Cholelithiasis after bariatric surgery, incidence, and prophylaxis: randomized controlled trial. Surg Endosc. 2020 Dec;34(12):5331-5337. doi: 10.1007/s00464-019-07323-7. Epub 2019 Dec 19. PMID 31858245
- [Background] Neuberg M, Blanchet MC, Gignoux B, Frering V. Long-Term Outcomes After One-Anastomosis Gastric Bypass (OAGB) in Morbidly Obese Patients. Obes Surg. 2020 Apr;30(4):1379-1384. doi: 10.1007/s11695-019-04287-4. PMID 31760607
- [Background] 3.Vural A, Goksu K, Kahraman AN et al. Increased gallstone formation after sleeve gastrectomy and the preventive role of ursodeoxycholic acid. Acta Gastroenterol Belg. 2020;83(1):33-38. 4. MAGOULIOTIS D.E., TASIOPOULOU V.S., SVOKOS A.A. et al.Ursodeoxycholic acid in the prevention of gall stone formation after bariatric surgery : A meta-analysis. Obese Sur., 2008, 27 : 3021-3030 5.MANATSATHIT W., LEELASINJAROEN P., AL-HAMID H., et al. The incidence of cholelithiasis after sleeve gastrectomy and its association with weight loss. A two-centre retrospective cohort study. Int Jpatients submitted to sleeve gastrectomy compared to normal subjects. Obes Surg., 2009, 19 : 1515-1521. 6. MELISSAS J., KOUKOURAKI S., ASKOXYLAKIS J., et al. Sleeve gastrectomy - Arestrictive procedure? Obes Surg., 2007, 17 : 57-62 7. LI V.K.M., PULIDO N., MARTINEZ-SUARTEZ P.et al. Symptomatic gallstones after sleeve gastrectomy. Surg Endosc., 2009, 23 : 2488-92. 8. Altieri, M. S., Yang, J., Nie, L., Docimo, S et al. Incidence of cholecystectomy after bariatric surgery. Surgery for Obesity and Related Diseases, (2018). 14(7), 992-996. 9. Morais M, Faria G, Preto J, et al. Gallstones and bariatric surgery: to treat or not to treat? World J Surg. 2016;40(12):2904-10. 10.Guzmán HM, Sepúlveda M, Rosso N. et al .Incidence and Risk Factors for Cholelithiasis After Bariatric Surgery [published correction appears in Obes Surg. 2019 May 28;:]. Obes Surg. 2019;29(7):2110-2114. doi:10.1007/s11695-019-03760-4. 11. Sioka E, Zacharoulis D, Zachari E et al. Complicated gallstones after laparoscopic sleeve gastrectomy. J Obes, 2014. 468203.